CLINICAL TRIAL: NCT00289354
Title: Randomized, Double Blinded, Placebo Controlled, Study to Evaluate Improvements in Glycemic Control, Lipid Levels, Quality of Life and Healthcare Costs After Daily Administration of Chromium Picolinate and Biotin in Patients With T2DM
Brief Title: Efficacy and Safety Study of Chromium Picolinate + Biotin on Glucose and Cholesterol Control in T2DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutrition 21, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N 21 CPB-02003
Record Dates: First submitted 2006-02-07; First posted 2006-02-09 (Estimated); Last update posted 2006-02-09 (Estimated); Status verified 2006-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: chromium; chromium picolinate; type 2 diabetes mellitus; HbA1c; hyperglycemia; cholesterol
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia | interventions — picolinic acid; Biotin

INTERVENTIONS:
Drug: Chromium Picolinate (600 mcg Cr) + biotin (2 mg)

SUMMARY:
To evaluate the effect of the combination of chromium picolinate (600 μg Cr) + biotin (2 mg) versus placebo on glycosylated hemoglobin (HbA1c), lipid profiles (Total-C, HDL-C, LDL-C, TGs, TG/HDL ratio, etc), and pharmacoeconomic outcomes as measured at the Baseline Visit and 90 days later at the Final Visit. Secondarily, to measure the effect of chromium picolinate (600 μg Cr) + biotin (2 mg) versus placebo on patient quality of life, fasting and post-prandial blood sugar levels, fasting insulin, and anti-hyperglycemic medication usage.

DETAILED DESCRIPTION:
There will be an Initial Pre-Screening Contact, two office visits (Baseline and Final), and two mid-study phone contacts with the subject during the course of the study. Volunteers will take either chromium picolinate (600 μg Cr) + biotin (2 mg) (n=400) or placebo (n=200) once daily just prior to the morning meal for 90 days. Assessments for glycosylated hemoglobin, lipid profiles, and quality of life will be taken at the Baseline Visit. After 90 days another set of assessments will be taken at the Final Visit for comparison with the baseline values. All subjects will under go a brief physical exam, a medical history assessment, and a comprehensive concomitant medications assessment as well as provide blood and urine samples at the baseline and final visits to ensure subject safety is maintained. The subject will be contacted, by a central call center, between visits at Day 30 and Day 60 to ensure study compliance by reminding the subject to take all doses of study product, perform the daily blood glucose monitoring, and complete the study diary daily.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of type 2 diabetes > 12 months.
2. Male and female between the ages of 18 and 70 years, inclusive.
3. HbA1c > 7.0%.
4. Subject must be receiving an anti-hyperglycemic medication. Medication dosage must be stable for at least 60 days prior to entering trial. Insulin usage must be for rescue purposes only. Rescue insulin use may not be more than once per week.
5. Subjects with a body mass index (BMI) >/= 25 and < 35.
6. Subject must be ambulatory.
7. Willing to perform self-administered blood glucose monitoring.
8. Willing to complete all study related requirements.
9. Subject will provide written consent to participate in the trial and this consent must be given voluntarily.

Exclusion Criteria:

1. Diagnosis of type 1 diabetes.
2. Hypoglycemic event requiring EMS intervention within 12 months.
3. Diabetic Ketoacidosis (DKA) within 12 months.
4. Subjects taking any supplement containing chromium picolinate within the last 90 days prior to enrollment.
5. Subjects taking a supplement or multivitamin containing any other form of chromium > 120 mcg/daily within the last 30 days prior to enrollment.
6. Creatinine > 2.0 x ULN; AST or ALT > 2.0 x ULN; Total Bilirubin > 1.5 x ULN
7. COPD, CHF, Angina, HTN, MI, or any other CVD requiring hospitalization within 12 months.
8. History of cerebrovascular accident (CVA), pulmonary embolism (PE), or an unresolved deep vein thrombosis (DVT).
9. History of CABG, PTCA, or any other reperfusion therapy within 12 months.
10. Seated systolic BP > 160 mmHg.
11. Morbid obesity.
12. Any psychiatric or mental health issue that would prevent the subject from completing the study. (e.g. Severe depression, schizophrenia, high suicide risk, bi-polar disorder, dementia, substance abuse, etc,)
13. History of any serious immunosuppressive disorder or current immunosuppressive therapy.
14. Female subjects who are pregnant or nursing, or are planning on becoming pregnant during the study.
15. Any illness or complication factor that, in the opinion of the investigator, would jeopardize the subject's health or well being by participating in the study or would interfere with the subject successfully completing the study.
16. Current diagnosis of any uncontrolled metabolic disease that would affect carbohydrate or glucose metabolism other than type 2 diabetes. (e.g. hyper or hypothyroidism). (NOTE: Subject's condition must be stable for > 12 months with no medication changes within the last 12 months preceding enrollment. Subject's TSH must be within range of normality at the time of enrollment to qualify).
17. Current participation in any other clinical research trial for any product or device, or participation in said clinical trials within 30 days prior to enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2003-03; Study Completion 2005-11

PRIMARY OUTCOMES:
HbA1c: Baseline and Final Visits
Lipid Panels (Total-C, HDL, LDL, LDL, VLDL, lipid ratios, etc)Baseline and Final Visits
Pharmacoeconomic outcomes (as deduced by changes in HbA1c)

SECONDARY OUTCOMES:
Fasting Plasma Glucose: Baseline and Final Visits
Fasting Insulin: Baseline and Final Visits
HOMA-IR and HOMA-BCF: Baseline and Final Visits
Quality of Life: Baseline and Final Visits
Post Prandial Glucose: Diary recordings of post meal values, 90 day continuous.
Change in Rx Antihyperglycemic agents: Assessed at baseline and compared to final visit.
HAMD-29: Change in depression/mood status; measured at baseline and final at a subset of two research centers. (n~30).
ANCOVAs: Treatment outcomes based on treatment group compared to gender, ethnicity, age, co-morbidities, Rx medications, glycemic states at entrance, lipid status at entrance.

CONTACTS AND LOCATIONS:
Overall Officials: Manley R Finch, Study Director — Nutrition 21, Inc.; Cesar Albarracin, MD, Principal Investigator — Alpha Therapy Center

REFERENCES:
- [Derived] Albarracin C, Fuqua B, Geohas J, Juturu V, Finch MR, Komorowski JR. Combination of chromium and biotin improves coronary risk factors in hypercholesterolemic type 2 diabetes mellitus: a placebo-controlled, double-blind randomized clinical trial. J Cardiometab Syndr. 2007 Spring;2(2):91-7. doi: 10.1111/j.1559-4564.2007.06366.x. PMID 17684468